CLINICAL TRIAL: NCT01022723
Title: Clinical Validation of a Microfluidic Device for Isolation and Molecular Characterization of Circulating Tumor Cells
Acronym: CTC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); National University of Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: CTC_ver2_081109
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Cancer
Keywords: Circulating tumor cells; metastasis; cancer; cell isolation; mircofludics; cell detection
MeSH Terms: conditions — Neoplasms; Neoplastic Cells, Circulating; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating Tumor Cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Lung Cancer patients: Lung Cancer (particular focus on non smokers with adenocarcinoma)
- Patients with Nasopharyneal carcinoma: Patients with Nasopharyneal carcinoma
- Breast Cancer patients: Breast cancer patients
- Prostate Cancer patients: Prostate cancer patients
- Colorectal Cancer patients: Colorectal cancer patients
- Gastric Cancer patients: Gastric cancer patients

SUMMARY:
To evaluate the efficiency of a microdevice for circulating tumor cells isolation and to correlate the circulating titre with response and progression.

DETAILED DESCRIPTION:
* Validate the clinical use of a mircofluidic device to capture circulating timor cells from a broad range of tumor types
* Characterize and identify these circulating tumor cells and demostrate cell viability with this capture method
* Apply this technology in clinically relevant settings and correlate to response to treatment and disease progression
* Elucidate predictive and pharmacodynamic biomarkers in the context of early phase trials of novel therapeutics

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed metastatic disease planned for palliative chemotherapy
* Tumor types as specified: non smokers with lung adenocarcinoma, undifferentiated EBV-ISH positive nasopharyneal carcinoma, breast cancer, colorectal cancer, prostate cancer, gastric cancer
* Informed consent given for the purposes of blood sampling for this study
* Measurable disease by RECIST criteria of at least 1cm is preferred but not a sine qua non for study accrual

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the following cancers:
  Lung Cancer Nasopharyneal carcinoma Breast cancer Prostate cancer Colorectal cancer Gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 817 (Estimated)
Dates: Start 2009-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The validation of the clinical use of a microfluidic device to capture circulating tumor cells (CTC) from a broad range of tumor types | 3 years

SECONDARY OUTCOMES:
Characteristics and viability of the CTC with this capture method | 3 years
Clinical application of this capture method with the study of CTC titre correlation to treatment outcome | 6 years
Study of predictive and pharmacodynamic biomarkers of the CTC in the context of early phase trials of novel therapeutics | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Teck Lim, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore